CLINICAL TRIAL: NCT06003712
Title: Exploring the Effects of a Mindfulness-Based Intervention on Physiologic and Quality of Life Markers in Individuals With Spinal Cord Injury (SCI): A Pre-post Test Design
Brief Title: Exploring the Effect of Mindfulness on Quality of Life (QoL) in Spinal Cord Injury (SCI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eduard Tiozzo, PhD, Principal Investigator, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230705
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Quality of Life
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Exercise Group (Experimental): Subjects will participate in a one-month mindfulness breathing-exercise program
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Participants will engage in a 10-15 minute mindfulness exercise three times weekly for one month. This mindfulness exercise utilizes guided attention on the breath through an instructional video, aiming to cultivate calmness and alleviate stress.

SUMMARY:
The purpose of this study is to determine if practicing mindfulness breathing exercises has an effect on the overall health of persons with SCI

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18-70 who are living with spinal cord injury
* C5 to the T10 levels
* Self-reported American Spinal Cord Injury Association (ASIA) Impairment Scale (AIS) A-D
* Eligible participants must be able to understand and provide consent, be in good health operationalized as free from acute treatable illness, pressure injury, and cardiovascular disease.

Exclusion Criteria:

* Participants taking medications that alter chronotropic and pressor responses will be excluded.
* Pregnant women will not be eligible to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Heart rate | baseline, 1 month
  heart rate will be collected in 5 minute intervals before, during and after the mindfulness sessions on 2 separate visits: baseline and post intervention visits. Heart rate will be recorded in beats per minute
Change in blood pressure | baseline, 1 month
  Blood pressure (BP) will be collected in 5 minute intervals before, during and after the mindfulness sessions on 2 separate visits: baseline and post intervention visits. BP will be collected as systolic over diastolic in mmHg units
Change in metabolism as measured by maximum oxygen consumption (VO2) | baseline, 1 month
  Metabolism as determined by oxygen consumption (VO2) will be collected in 5 minute intervals before, during and after the mindfulness sessions on 2 separate visits: baseline and post intervention visits. VO2 is collected as mL/kg/min
Change in metabolism as measured by ventilation (VE) | baseline, 1 month
  Metabolism as determined by oxygen consumption (VE) will be collected in 5 minute intervals before, during and after the mindfulness sessions on 2 separate visits: baseline and post intervention visits. VE is measured in L/min

SECONDARY OUTCOMES:
Change in Quality of Life (QoL) as measured by Quality Index Spinal Cord Injury Version III | baseline, 1 month
  A composite score will be obtained to assess change in QoL using a six-point Likert scale. Scores for satisfaction section range from "1- very satisfied" to "6-very dissatisfied". On the important section scoring ranges from "1-very important" to "6- very unimportant"

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Tiozzo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami - Miami Project to Cure Paralysis, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No